CLINICAL TRIAL: NCT05044156
Title: Investigation of the Relationship Between Salivary Histatine-5 Level and Vaginal Candidiasis in Women
Status: Completed | Type: Observational
Sponsor: Usak State Hospital (Other)
Responsible Party: Principal Investigator, Irem Senyuva, M.D, Obstetrics and Gynecology, Usak State Hospital
Other Study IDs: Usak State Hospital
Record Dates: First submitted 2021-09-04; First posted 2021-09-14 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Vaginal Infection; Candidiasis
MeSH Terms: conditions — Vaginitis; Candidiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: vaginal candidiasis
  Interventions: Other: salivary sample
- Control group: healty women
  Interventions: Other: salivary sample

INTERVENTIONS:
Other: salivary sample — salivary sample

SUMMARY:
The low Histatine-5 (HST-5) level of the saliva can lead to vaginal candidiasis. Because HST-5 level in the saliva can effect vaginal Ph, flora and local defence mechanisms.

Histatine-5 is secreted in the parotis and submandibular glands. İt riches histidine amino ascid and have antifungal activity. Salivary proteins and their plasma levels were found as similar in the literature.

DETAILED DESCRIPTION:
Women with regularly menstrual cycle will enroll in the study than will separate two groups:

Study group: women with vaginal candidiasis ( diagnosed by clinic and lab.)

Control group: women ( not have any vaginal infections candida and others)

Saliva samples will be taken from two groups than HST-5 level will be analyzed. Finally HST-5 levels of the two groups will be compared .

Women with diabetes, immun deficiency, pregnancy, virgin, menopausal period , premature ovarian failure will be excluded.

ELIGIBILITY:
Inclusion Criteria: women with regularly menstrual cycle , diagnosed candidal vaginosis and not have any vaginal infection.

-

Exclusion Criteria: diabetes, immun deficiency, menopause, premature ovarian failure, pregnancy, virgin

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: women with regularly menstrual cycle, diagnosed candidal vaginosis and not have any vaginal infection.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
SALIVARY HISTATINE-5 LEVEL IN THE WOMEN WITH VAGINAL CANDIDIASIS | 1 month
  we done salivary protein electrophoresis( as a small sample group ; consist of vaginal candidiasis and control patients) and Hst5 protein band was seen

SECONDARY OUTCOMES:
SALIVARY HISTATINE-5 LEVEL IN THE WOMEN WITH VAGINAL CANDIDIASIS | 2 month
  We found , low salivary Hst5 levels in women with vaginal candidiasis than control group (p=0.001)

CONTACTS AND LOCATIONS:
Overall Officials: İREM ŞENYUVA, M.D, Principal Investigator — USAK TRAINING AND RESEARCH HOSPITAL
Locations (1):
- İrem Şenyuva, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khurshid Z, Najeeb S, Mali M, Moin SF, Raza SQ, Zohaib S, Sefat F, Zafar MS. Histatin peptides: Pharmacological functions and their applications in dentistry. Saudi Pharm J. 2017 Jan;25(1):25-31. doi: 10.1016/j.jsps.2016.04.027. Epub 2016 May 4. PMID 28223859
- [Background] Loo JA, Yan W, Ramachandran P, Wong DT. Comparative human salivary and plasma proteomes. J Dent Res. 2010 Oct;89(10):1016-23. doi: 10.1177/0022034510380414. Epub 2010 Aug 25. PMID 20739693
- [Background] Liao H, Liu S, Wang H, Su H, Liu Z. Efficacy of Histatin5 in a murine model of vulvovaginal candidiasis caused by Candida albicans. Pathog Dis. 2017 Aug 31;75(6). doi: 10.1093/femspd/ftx072. PMID 28645176